CLINICAL TRIAL: NCT06681753
Title: Associate Professor Öznur Tiryaki Sakarya University
Brief Title: The Effect of Breastfeeding Support Education on Midwifery Profession Perception and Belonging
Acronym: Midwifery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, associate professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E-61923333-050.99-27167
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Breastfeeding
Keywords: Breast milk; Midwifery; Belonging; Profession
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Pretest-posttest matched control group quasi-experimental
Who Masked: Participant
Masking Description: Sampling Inclusion Criteria:
  * Being a senior student in the SAU Faculty of Health Sciences, Midwifery Department
  * The student agrees to participate in the study
  Sampling Exclusion Criteria:
  * The student does not agree to participate in the study
  * Being a 1st, 2nd or 3rd year student in the SAU Faculty of Health Sciences, Midwifery Department
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Breastfeeding Consultancy and Baby Friendly Hospital Training Program (Experimental): The project consultant (PT) who is a Breastfeeding Consultant and National Baby Friendly Hospital evaluator and a nurse working in the Neonatal Intensive Care Unit and who participated in the Breastfeeding Consultancy and Baby Friendly Hospital Training Program of the Ministry of Health, will provide 6 hours of theoretical and 2 hours of practical training on Breastfeeding and Breastfeeding support. The training content will include the following topics: Breastfeeding Status in Turkey and the World, Effective Communication and Consultancy Skills, Composition of Breast Milk, Lactation and Relaxation, Breastfeeding Positions, Feeding of Babies with Special Conditions, and Benefits of Breastfeeding.
  Interventions: Other: Experimental
- Control (No Intervention)

INTERVENTIONS:
Other: Experimental — No training will be planned for the Control Group, and their undergraduate education will be included in the study. After the study data is collected and the study is concluded, the control group will be given breastfeeding support training from the intervention group.
  Other Names: Control
  Arms: the Breastfeeding Consultancy and Baby Friendly Hospital Training Program

SUMMARY:
The study was planned to provide knowledge and skills regarding breast milk and breastfeeding to midwifery students who will provide breast milk and breastfeeding consultancy to women and the society during pregnancy, birth and postpartum period after graduation, and to positively develop their professional affiliation and perception of the profession.

In this context, the following hypotheses will be tested in the study:

H0: Breastfeeding support education has no effect on the professional affiliation and perception of the profession of intern midwifery students.

H1: Breastfeeding support education increases the breastfeeding and breast milk knowledge and skills of intern midwifery students.

H2: Breastfeeding support education increases the professional affiliation of intern midwifery students.

H3: Breastfeeding support education positively develops the professional perception of intern midwifery students

DETAILED DESCRIPTION:
The universe of the study will consist of all students studying in the Department of Midwifery at SAU Faculty of Health Sciences, and the sample will consist of senior midwifery students. In order to determine the sample size, a power analysis will be conducted using the G*Power (v3.1.7) program. The aim of the study was to evaluate the differences in the mean knowledge level scores between the groups. The effect width value was taken as 0.70 as the method used in cases where it is not known how many units of difference are significant between the groups. The effect width value of 0.20 is very high, 0.50 is at a medium level, and 0.80 gives results under the maximum acceptance limit. As the power of the study increases, it means that the measurement is more sensitive in finding the difference. The power is expected to be 0.80 and above. In the case of a Type 1 error probability (α) of 0.05 (95% confidence interval), a power level of 80%, and an effect width value of 0.70, the study will be planned with a total of 68 students, 34 students for each group. Considering the possibility of data collection forms being incomplete and empty, 10% of the sample size (37 for each group, totaling 74 students who meet the inclusion criteria) will be included in the study. When the desired number is reached for each group during the study process, the power of the study will be calculated again (post hoc).

Criteria for Inclusion in the Sample:

* Being a senior student in the SAU Faculty of Health Sciences, Midwifery Department
* The student agrees to participate in the study

Criteria for Exclusion from the Sample:

* The student does not agree to participate in the study
* Being a 1st, 2nd and 3rd year student in the SAU Faculty of Health Sciences, Midwifery Department Data Collection Tools: Data will be collected using the Demographic Information Form containing the sociodemographic characteristics of the participants, the Breast Milk and Breastfeeding Questionnaire prepared by the researchers in line with the literature, the Midwifery Belonging Scale and the Midwifery Profession Perception Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being a senior student in the SAU Faculty of Health Sciences, Midwifery Department
* The student agrees to participate in the study

Exclusion Criteria:

* The student does not agree to participate in the study
* Being a 1st, 2nd or 3rd year student in the SAU Faculty of Health Sciences, Midwifery Department

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
To provide intern midwifery students with breastfeeding consultancy skills. | 12 WEEKS
  scale scores will be evaluated
To ensure that they embrace the midwifery profession and gain a sense of belonging. | 12 WEEKS
  scale scores will be evaluated

SECONDARY OUTCOMES:
To create awareness so that they can better perceive the midwifery profession by realizing the duties, authorities and responsibilities of the profession. | 12 WEEKS
  scale scores will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Öznur Tiryaki, PhDr, Study Chair — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No